CLINICAL TRIAL: NCT06991166
Title: OBWELL: Evaluating the Effectiveness of an Innovative Psychotherapeutic Intervention to Treat Postpartum Depression Among High-Risk Mothers
Brief Title: OBWELL: Innovative Psychotherapeutic Intervention to Treat Postpartum Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Collaborators: New Jersey Health Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro2024-0204
Record Dates: First submitted 2025-05-19; First posted 2025-05-26 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Post Partum Depression
Keywords: Post Partum Depression; Cognitive behavioral therapy; interpersonal therapy; psychotherapy; NICU
MeSH Terms: conditions — Depression, Postpartum | interventions — Cognitive Behavioral Therapy; Psychotherapy, Group; Telemedicine; adenylate isopentenyltransferase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4-week Cognitive behavioral therapy (CBT) psychotherapy group/telehealth intervention (Experimental): After the first 4-week of CBT intervention , participants will be administered the Peri-Intervention (Week 4) Assessment - which consists of the EPDS, Social Determinants of Health, and the Risk Factor questionnaire - and then "cross-over" to the second 4-week of IPT intervention.
  Interventions: Behavioral: Cognitive behavioral therapy (CBT) psychotherapy group/telehealth; Behavioral: Interpersonal therapy (IPT) psychotherapy group/telehealth
- 4-week interpersonal therapy (IPT) psychotherapy group/telehealth intervention (Experimental): After the first 4-week of IPT intervention , participants will be administered the Peri-Intervention (Week 4) Assessment - which consists of the EPDS, Social Determinants of Health, and the Risk Factor questionnaire - and then "cross-over" to the second 4-week of CBT intervention.
  Interventions: Behavioral: Cognitive behavioral therapy (CBT) psychotherapy group/telehealth; Behavioral: Interpersonal therapy (IPT) psychotherapy group/telehealth

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy (CBT) psychotherapy group/telehealth — Type of psychotherapy. CBT focuses on identifying and changing unhelpful beliefs and behavioral patterns that lead to negative emotions (e.g., depression, anxiety, grief, shame) in order to break the emotion-thought-behavior cycle
Behavioral: Interpersonal therapy (IPT) psychotherapy group/telehealth — Type of psychotherapy. IPT focuses on improving interpersonal communication and deficits, processing grief, and role transitions

SUMMARY:
Postpartum Depression (PPD) is defined as depression that occurs after childbirth, with intense symptoms that last longer than "baby blues". PPD differs greatly from "baby blues", a term used to describe the typical sadness, worry and tiredness that women experience after childbirth, which often resolves within a week or two on its own. The symptoms of PPD interfere with many aspects of daily living and can have unhealthy short-term and long-term outcomes, both for the mother and baby.

One-third of women in the U.S. with PPD are identified in clinical settings, yet only half of those begin psychotherapy treatment. Unfortunately, mothers whose newborns are in the Neonatal Intensive Care Unit (NICU) are at high risk for developing PPD, necessitating early identification and evidence-based treatment. Cognitive behavioral therapy (CBT) and interpersonal therapy (IPT) are the two most effective psychotherapy treatments for PPD, yet no randomized controlled clinical trials were found that directly compared the two types of treatment or determined whether combining the two approaches is more helpful for PPD than either approach alone.

This clinical trial aims to compare the effectiveness of a 4-week intervention of either CBT or IPT for PPD in NICU mothers and to determine whether a sequential 8-week intervention (IPT then CBT, or CBT then IPT) is more beneficial.

ELIGIBILITY:
Inclusion Criteria:

* Mother of NICU infant
* Older than age 18
* English-speaking
* Gave birth more than 24 hours ago and less than 12 months prior to enrollment
* Depression as assessed by:

Current/Prior diagnosis of Major Depressive Disorder OR EPDS score above 10 OR EPDS score below 10 AND Endorsement of "sometimes" or "often" on item #10 on the EPDS* ("I have had thoughts of harming myself")

Exclusion Criteria:

* A diagnosis of Substance Dependency or Substance Use
* Acute suicidal or infanticidal ideation
* Current psychosis
* Medical history of cognitive impairment
* Infant death of current NICU admission
* Marked non-compliance with intervention (e.g, non-attendance of more than one session during a 4-week intervention or failure to complete study assessments),
* Are in medical treatment that would prevent participation (i.e., medical treatment that requires inpatient hospitalization and thus would prevent participation of study visits.)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Mothers with babies at the NICU
Enrollment: 72 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Post Partum Depression post initial psychotherapy | At 4 weeks
  Quantitative assessment of treatment effectiveness in reducing PPD symptoms will be conducted with the Edinburgh Postnatal Depression Scale (EPDS), a 10-item validated self-report scale. Total scores on the EPDS range from 0 to 30, with scores 13 and above indicating depressive illness, or a high risk of developing a depressive disorder. The measures will be administered at the following timepoints:
  Week 0 Baseline: At study entry prior to starting group psychotherapy in the Outpatient Behavioral Health practice Week 4: After completing the first 4-week intervention of the two-intervention sequence, prior to "crossing over"

SECONDARY OUTCOMES:
Postpartum Depression after both types of psychotherapy | At 8 weeks
  Quantitative assessment of treatment effectiveness in reducing PPD symptoms will be conducted with the Edinburgh Postnatal Depression Scale (EPDS), a 10-item validated self-report scale. Total scores on the EPDS range from 0 to 30, with scores 13 and above indicating depressive illness, or a high risk of developing a depressive disorder. The measure will be administered at Week 8: After completing the second 4-week intervention and completing the entire 8-week two-intervention sequence.
Postpartum Depression at follow up | At 6 months
  Quantitative assessment of treatment effectiveness in reducing PPD symptoms will be conducted with the Edinburgh Postnatal Depression Scale (EPDS), a 10-item validated self-report scale. Total scores on the EPDS range from 0 to 30, with scores 13 and above indicating depressive illness, or a high risk of developing a depressive disorder. The measure will be administered at 6 months post enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Yeraz Markarian, PhD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack University Medical Center, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saharoy R, Potdukhe A, Wanjari M, Taksande AB. Postpartum Depression and Maternal Care: Exploring the Complex Effects on Mothers and Infants. Cureus. 2023 Jul 4;15(7):e41381. doi: 10.7759/cureus.41381. eCollection 2023 Jul. PMID 37546054
- [Background] Cox EQ, Sowa NA, Meltzer-Brody SE, Gaynes BN. The Perinatal Depression Treatment Cascade: Baby Steps Toward Improving Outcomes. J Clin Psychiatry. 2016 Sep;77(9):1189-1200. doi: 10.4088/JCP.15r10174. PMID 27780317
- [Background] Wyatt T, Shreffler KM, Ciciolla L. Neonatal intensive care unit admission and maternal postpartum depression. J Reprod Infant Psychol. 2019 Jul;37(3):267-276. doi: 10.1080/02646838.2018.1548756. Epub 2018 Nov 19. PMID 30450956
- [Background] Bonacquisti A, Geller PA, Patterson CA. Maternal depression, anxiety, stress, and maternal-infant attachment in the neonatal intensive care unit. J Reprod Infant Psychol. 2020 Jul;38(3):297-310. doi: 10.1080/02646838.2019.1695041. Epub 2019 Dec 4. PMID 31795733
- [Background] Stamou G, Garcia-Palacios A, Botella C. Cognitive-Behavioural therapy and interpersonal psychotherapy for the treatment of post-natal depression: a narrative review. BMC Psychol. 2018 Jun 18;6(1):28. doi: 10.1186/s40359-018-0240-5. PMID 29914574
- [Background] Stuart S, Koleva H. Psychological treatments for perinatal depression. Best Pract Res Clin Obstet Gynaecol. 2014 Jan;28(1):61-70. doi: 10.1016/j.bpobgyn.2013.09.004. Epub 2013 Oct 7. PMID 24269903
- [Background] Burger M, Hoosain M, Einspieler C, Unger M, Niehaus D. Maternal perinatal mental health and infant and toddler neurodevelopment - Evidence from low and middle-income countries. A systematic review. J Affect Disord. 2020 May 1;268:158-172. doi: 10.1016/j.jad.2020.03.023. Epub 2020 Mar 6. PMID 32174474
- [Background] Stevenson MD, Scope A, Sutcliffe PA, Booth A, Slade P, Parry G, Saxon D, Kalthenthaler E; group cognitive behavioural therapy for postnatal depression advisory group. Group cognitive behavioural therapy for postnatal depression: a systematic review of clinical effectiveness, cost-effectiveness and value of information analyses. Health Technol Assess. 2010 Sep;14(44):1-107, iii-iv. doi: 10.3310/hta14440. PMID 20863477
- [Background] Klier CM, Muzik M, Rosenblum KL, Lenz G. Interpersonal psychotherapy adapted for the group setting in the treatment of postpartum depression. J Psychother Pract Res. 2001 Spring;10(2):124-31. PMID 11264336
- [Background] Beck, J.S.(2021) Cognitive Behavior Therapy : Basics and Beyond, Third Edition, NY: Guilford Press